CLINICAL TRIAL: NCT02013505
Title: A Validated Educational Video Intervention Improves the Quality of Bowel Preparation for Colonoscopy.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study expired; Investigator left facility.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1203774
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Bowel Dysfunction
Keywords: Colonoscopy
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Instructions printed on a paper. (No Intervention): There will be no intervention.
- Paper and video instructions (Experimental): .Instructions printed on paper and a educational video.
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — An educational video was developed based on the current paper instructions for bowel preparation. The video included a physician explaining the process, using more images and short clip videos of the example. The script of the video was approved by the patient education department of the University Hospital and language adjusted to 6th grade level.
  Arms: Paper and video instructions

SUMMARY:
The investigators hypothesised that a video based patient education will help patients understand the process of colon cleansing prior to a colonoscopy procedure and hence will result in clean colons that will may help physician perform a better quality examination.

DETAILED DESCRIPTION:
After obtaining consent over phone, the investigators randomly assigned assigned participants to receive either the standard paper based instructions or receive an educational video in addition to the standard paper based instruction. Physicians performing the procedure were blinded to this assignment. The investigators obtained information relating to the cleanliness of the colon as noted during the colonoscopy examination. The investigators obtained this information from the colonoscopy reports. The investigators also obtained information regarding colon polyps,wanting to see if there is any difference in the number of patients in whom adenomatous polyps were detected.

Outcome measures:

Primary Out come:

1.Quality of bowel preparation

Secondary outcome:

1. Adenoma detection rate
2. Rate of incomplete procedures due to poor bowel prep.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Subjects who have the ability to give consent
3. Subjects who are scheduled for colonoscopy as out patient
4. Subjects consenting to participate in the study
5. Subjects who are able to read and understand English

Exclusion Criteria:

1. < 18 years age
2. Subjects from whom consent cannot be obtained for any reason.
3. Subjects who are scheduled for colonoscopy as in patient
4. Subjects who are scheduled for colonoscopy within a time period or a situation where the educational material cannot be properly delivered to the study participant.
5. Subjects who are advised to undergo bowel prep for more than one day.
6. Subjects undergoing bowel prep with medications other than Colyte.
7. Subjects who do not have access to equipment to watch the video (TV/CD player)
8. Pregnant patients
9. Prisoners
10. Subjects who are not able to read or understand English.

(j)Subjects who had bowel resection surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | At the time of colonoscopy
  Quality of bowel preparation at the time when the colonoscopy procedure is performed as reported by the physician performing the colonoscopy.

SECONDARY OUTCOMES:
Adenoma detection rate | At time of colonoscopy
  Number of patients undergoing screening colonoscopy for average risk in whom an adenoma was detected.

CONTACTS AND LOCATIONS:
Overall Officials: Dilip Bearelly, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No